CLINICAL TRIAL: NCT03614234
Title: Open Label Extension Study to Evaluate the Long-term Safety and Efficacy of 2 mg/kg Pegunigalsidase Alfa (PRX-102) Administered by Intravenous Infusion Every 4 Weeks in Adult Patients With Fabry Disease
Brief Title: Open Label Extension of 2 mg/kg Pegunigalsidase Alfa (PRX-102) Every 4 Weeks in Adult Fabry Disease Patients
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLI-06657AA1-03
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Fabry Disease
Keywords: Glomerular filtration rate; Proteinuria; PRX-102; pegunigalsidase alfa; Fabry disease
MeSH Terms: conditions — Fabry Disease; Proteinuria

STUDY DESIGN:
Intervention Model Description: Open-label extension study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental open label (Experimental): Pegunigalsidase alfa
  Interventions: Drug: pegunigalsidase alfa

INTERVENTIONS:
Drug: pegunigalsidase alfa — Recombinant human alpha galactosidase A
  Other Names: PRX-102

SUMMARY:
The objective of CLI-06657AA1-03 (formerly PB-102-F51) is to evaluate the long-term safety, tolerability, and efficacy of 2 mg/kg pegunigalsidase alfa administered intravenously every four weeks in adult Fabry patients who have successfully completed PB-102-F50.

DETAILED DESCRIPTION:
This is an open-label study to assess the long-term safety and efficacy of pegunigalsidase alfa treatment of 2.0 mg/kg administered intravenously every 4 weeks. The duration of treatment will be until pegunigalsidase alfa is commercially available to the patient, or at the discretion of the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of study PB-102-F50.
2. The patient signs informed consent.
3. Female patients and male patients whose co-partners are of child-bearing potential agree to use a medically accepted, effective contraception method. These include combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal) supplemented with a barrier method (preferably male condom), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable) supplemented with a barrier method (preferably male condom), intrauterine device (IUD), intrauterine hormone-releasing system (IUS), bilateral tubal occlusion, vasectomised partner, or sexual abstinence. Contraception should be used for 2 weeks after treatment termination.

Exclusion Criteria:

Presence of any medical, emotional, behavioral, or psychological condition that, in the judgment of the Investigator, would interfere with patient compliance with the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-11-13 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment-related adverse events | Throughout the study, 364 weeks
  CTCAE v4.03

SECONDARY OUTCOMES:
Kidney function 1 | Every 6 months throughout the duration of the study, 364 weeks
  Estimated glomerular filtration rate (eGFRCKD-EPI)
Cardiac assessment | Once a year throughout the study at weeks 52, 104, 152, 200, 256, 312 and end of study week 364
  Left Ventricular Mass Index (g/m2) by echocardiogram and cardiac function stress test
Biomarkers for Fabry disease | Every 6 months throughout the duration of the study, 364 weeks
  Plasma Lyso-Gb3 and Gb3
Kidney function 2 | Every 6 months throughout the duration of the study, 364 weeks
  Protein/Creatinine ratio (UPCR), spot urine test
Clinical assessment | Every four weeks throughout the duration of the study, 364 weeks
  Record of pain medication and pre-medication use
Pain assessment | Every 6 months throughout the duration of the study, 364 weeks
  Short form Brief Pain Inventory (BPI)
Symptom assessment | Once a year throughout the study at weeks 52, 104, 152, 200, 256, 312 and end of study week 364
  Mainz Severity Score Index (MSSI)
Quality of life assessment | Every 6 months throughout the duration of the study, 364 weeks
  Quality of life (EQ-5D-5L)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (7):
  - UAB Medicine, Birmingham, Alabama
  - Emory University School of Medicine, Atlanta, Georgia
  - University of Iowa Hospitals and Clinica, Iowa City, Iowa
  - Infusion Associates, Grand Rapids, Michigan
  - Renal Disease Research Institute, LLC, Dallas, Texas
  - University of Utah Hospitals & Clinics, Salt Lake City, Utah
  - O & O Alpan, Fairfax, Virginia
- UZ Antwerpen, Edegem, Belgium
- Fakultní poliklinika Všeobecné fakultní nemocnice v Praze, Prague, Czechia
- Medical Endocrinology PE 2132, Rigshospitalet, Copenhagen, Denmark
- Azienda Ospedaliera Universitaria "Federico II", Napoli, Via Pansini, Italy
- Helse Bergen HF Haukeland Universitetssykehus, Bergen, Norway
- United Kingdom (2):
  - Addenbrooke's Hospital, Cambridge
  - The Royal Free Hospital, London